CLINICAL TRIAL: NCT04635943
Title: Randomized Phase IIA Clinical Trial to Evaluate the Efficacy of Ivermectin to Obtain Negative PCR Results in Patients With Early Phase COVID-19
Acronym: SAINT-PERU
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidad Peruana Cayetano Heredia (Other)
Collaborators: Barcelona Institute for Global Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EC-CNTEI-014-2020
Record Dates: First submitted 2020-11-09; First posted 2020-11-19 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-03

CONDITIONS: Covid19; Coronavirus Infection; SARS-CoV Infection
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Severe Acute Respiratory Syndrome | interventions — Ivermectin

STUDY DESIGN:
Intervention Model Description: SAINT-PERU is a triple-blinded, randomized, placebo-controlled trial with two parallel arms to evaluate the efficacy of one daily dose of ivermectin during three consecutive days, administered to patients with a positive PCR test for SARS-CoV-2 in a nasopharyngeal specimen, symptomatic for 96 hours or less, with non-severe COVID-19 disease at baseline, regardless of the presence of risk factors for progression to severity. The efficacy of the drug-based strategy to reduce or block transmission involves treating during early phases of infection, when viral replication is yet limited.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The Ivermectin presentation will be an oral drop solution in a flasks containing 5ml. The placebo presentation will also be an oral drop solution, undistinguishable from ivermectin, but without this device pharmaceutical ingredient. The pharmacist will prepare the treatment flasks (three 5ml flasks per participant), labelling them according to the randomization list in blocks of four (a, b) previously prepared by the epidemiologist, and according to the randomized treatment allocation previously notified by the principal investigator. The participant, investigator and outcomes assessor will be blinded to the study intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ivermectin (Active Comparator): Participants on this arm will receive orally one (1) daily dose of ivermectin 300 mcg/kg for three (3) consecutive days, starting at the enrolment visit.
  Interventions: Drug: Ivermectin
- Placebo (Placebo Comparator): Participants on this arm will receive orally one (1) daily dose of placebo for three (3) consecutive days, starting at the enrolment visit.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ivermectin — One daily dose of NOXAL-Ivermectin Oral Solution (6 mg/mL) at 300mcg/kg for three (3) consecutive days. A weight-equivalence table will be used to determine each participant´s dose (number of oral drops/day).
  Other Names: Noxal
  Arms: Ivermectin
Drug: Placebo — The placebo presentation will be an oral drop solution undistinguishable from ivermectin, but without this device pharmaceutical ingredient.
  Arms: Placebo

SUMMARY:
SAINT-PERU is a triple-blinded, randomized placebo-controlled trial with two parallel arms to evaluate the efficacy of ivermectin in negativizing nasopharyngeal PCR in patients with SARS-CoV-2 infection. The trial is conducted in two national hospitals at Lima-Peru.

DETAILED DESCRIPTION:
SAINT is a triple-blinded, randomized placebo-controlled trial with two parallel arms to evaluate the efficacy of ivermectin in negativizing nasopharyngeal PCR in patients with SARS-CoV-2 infection. The trial is conducted in two national hospitals at Lima-Peru.

The planned sample size is 186 SARS-CoV-2 PCR positive patients: 93 patients to treatment and 93 to the placebo group. Participants will be randomized to receive one dose of 300 mcg/kg ivermectin or placebo daily for three consecutive days. The epidemiologist will generate a list of correlative numbers, in randomized blocks of size 4, with the assignment to the treatment groups (a and b). The randomization list will be kept in an encrypted file accessible only to the trial statistician. This list will be handed directly to the pharmacist. Independently, the principal investigator will randomly assign the intervention (ivermectin) to one of the two groups (a or b) by tossing a coin, and will inform the pharmacist of the result of this process. The pharmacist will prepare and label the treatment vials according to the randomization list prepared by the epidemiologist and the treatment assignment given by the principal investigator. Eligible patients will be allocated in a 1:1 ratio using this randomization list.

Participants are expected to remain in the trial for a period of 21 days.

In the interests of public health and containing transmission of infection, follow-up visits will be conducted by the trial medical staff at the participant's home or at a hospital in case of hospitalization.

Follow-up visits will assess clinical and laboratory parameters of the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with COVID-19 typical symptoms (cough, fever, anosmia) present for not more than 96 hours.
2. 18 years or older.
3. No use of ivermectin prior to the study.
4. No known history of ivermectin allergy.
5. The patient can give his consent to take part in the study.
6. Not current use of CYP 3A4 or P-gp inhibitor drugs such as quinidine, amiodarone, diltiazem, spironolactone, verapamil, clarithromycin, erythromycin, itraconazole, ketoconazole, cyclosporine, tacrolimus, indinavir, ritonavir or cobicistat. Use of critical CYP3A4 substrate drugs such as warfarin.

Exclusion Criteria:

1. COVID-19 pneumonia

   * Diagnosed by the attending physician (oxygen saturation < 95% or lung crackles)
2. Positive pregnancy test for women of childbearing age*
3. Positive IgG against SARS-CoV-2 by rapid diagnostic test.
4. Negative SARS-CoV-2 PCR from a nasopharyngeal swab.

   * Women of child bearing age may participate if they use a safe contraceptive method for the entire period of the study. A woman is considered to not have childbearing capacity if she is post-menopausal (minimum of 2 years without menstruation) or has undergone surgical sterilization (at least one month before the study)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2020-08-29 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with a positive SARS-CoV-2 PCR. | 7 days post-treatment
  Proportion of patients with a positive SARS-CoV-2 PCR from a nasopharyngeal swab at day 7 post-treatment

SECONDARY OUTCOMES:
Mean viral load | Baseline and on days 4, 7, 14 and 21
  Change from baseline quantitative and semi-quantitative PCR in nasopharyngeal swab
Fever and cough progression | Up to and including day 21
  Proportion of patients with fever and cough at days 4, 7, 14 and 21 as well as proportion of patients progressing to severe disease or death during the trial
Seroconversion at day 21 | Up to and including day 21
  Proportion of participants with positive IgG at day 21
Proportion of drug-related adverse events | 7 days post treatment
  Proportion of drug-related adverse events
Levels of IgG, IgM and IgA | Up to and including day 21
Frequency of innate immune cells | Up to and including day 7
  Frequency (% over total PBMC) of innate immune cells (myeloid and plasmacytoid dendritic cells, NK cell, classical, intermediate and pro-inflammatory macrophages) measured in cryopreserved PBMC by flow cytometry
Frequency SARS-CoV-2-specific CD4+ T and and CD8+ T cells | Up to and including day 7
  Frequency of CD4+ T and CD8+ T cells (% over total CD4+T and CD8+ T) expressing any functional marker upon in vitro stimulation of PBMC with SARS-CoV-2 peptides, measured by flow cytometry
Results from cytokine Human Magnetic 30-Plex Panel | Up to and including day 21
  Concentration (all in pg/mL) of epidermal growth factor (EGF), fibroblast growth factor (FGF), granulocyte colony-stimulating factor (G-CSF), granulocyte-macrophage colony-stimulating factor (GM-CSF), hepatocyte growth factor (HGF), vascular endothelial growth factor (VEGF), tumour necrosis factor (TNF), interferon (IFN)-α, IFN-γ, interleukin (IL)-1RA, IL-1β, IL-2, IL-2R, IL-4, IL-5, IL-6, IL-7, IL-8, IL-10, IL-12(p40/p70), IL-13, IL-15, IL-17, IFN-γ induced protein (IP-10), monocyte chemoattractant protein (MCP-1), monokine induced by IFN-γ (MIG), macrophage inflammatory protein (MIP)-1α, MIP-1β in plasma measured by a Luminex assay using a commercially available kit (Cytokine Human Magnetic 30-Plex Panel from ThermoFisher)
Presence of intestinal helminths | Baseline and on day 14.
  Proportion and parasitic load of intestinal helminths by spontaneous sedimentation method.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Nacional Cayetano Heredia, Lima, Peru

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Garcia PJ, Mundaca H, Ugarte-Gil C, Leon P, Malaga G, Chaccour C, Carcamo CP. Randomized clinical trial to compare the efficacy of ivermectin versus placebo to negativize nasopharyngeal PCR in patients with early COVID-19 in Peru (SAINT-Peru): a structured summary of a study protocol for randomized controlled trial. Trials. 2021 Apr 9;22(1):262. doi: 10.1186/s13063-021-05236-2. PMID 33836826